CLINICAL TRIAL: NCT00096460
Title: Autologous Versus Non-Myeloablative Allogeneic Hematopoietic Stem Cell Transplantation (HSCT) for Patients With Chemosensitive Follicular Non-Hodgkin's Lymphoma Beyond First Complete Response or First Partial Response (BMT CTN #0202)
Brief Title: Autologous or Donor Stem Cell Transplantation in Treating Patients With Recurrent Non-Hodgkin's Lymphoma (BMT CTN 0202)
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: lower than anticipated accrual
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Blood and Marrow Transplant Clinical Trials Network (Network); National Cancer Institute (NCI) (NIH); National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMTCTN0202; U01HL069294 (NIH); BMT CTN 0202 (Other: Blood and Marrow Transplant Clinical Trials Network); 5U24CA076518 (NIH)
Record Dates: First submitted 2004-11-09; First posted 2004-11-10 (Estimated); Results first posted 2012-09-17 (Estimated); Last update posted 2023-01-05 (Actual); Status verified 2022-12

CONDITIONS: Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Cyclophosphamide; Rituximab; Filgrastim; Granulocyte Colony-Stimulating Factor; Drug Therapy; Radiotherapy; Etoposide; Carmustine; fludarabine; fludarabine phosphate; Transplantation, Homologous; Transplantation, Autologous; Tacrolimus; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Autologous Transplant (Active Comparator): Cyclophosphamide and Rituximab with Filgrastim conditioning and chemotherapy or radiation therapy prior to autologous Hematopoietic Stem Cell Transplant (HSCT). Rituximab maintenance therapy following HSCT.
  Interventions: Drug: Cyclophosphamide and Rituximab; Drug: Filgrastim; Radiation: Chemotherapy or Radiation therapy; Procedure: Autologous transplant; Drug: Rituximab maintenance therapy
- Allogeneic Transplant (Active Comparator): Non-myeloablative conditioning regimen followed by allogeneic Hematopoietic Stem Cell Transplant (HSCT). Graft-versus-Host Disease (GVHD) Prophylaxis therapy following HSCT.
  Interventions: Drug: Cyclophosphamide and Rituximab; Drug: Filgrastim; Drug: Non-myeloablative Conditioning regimen; Procedure: Allogeneic transplant; Drug: GVHD Prophylaxis

INTERVENTIONS:
Drug: Cyclophosphamide and Rituximab — Prior to undergoing HSCT, all patients will receive Cyclophosphamide 4 gm/m2 with Rituximab 375 mg/m2 x 2 doses and G-CSF support.
  Other Names: Cytoxan® and Rituxan
Drug: Filgrastim — Autologous HSCT patients will receive 10 mcg/kg/day and allogeneic HSCT patients will receive 5 mcg/kg/day subcutaneous (SQ) or intravenous (IV) starting 2 days after the initiation of Cyclophosphamide.
  Other Names: G-CSF
Radiation: Chemotherapy or Radiation therapy — Chemotherapy - BCNU 15 mg/kg IV x 1 dose to be administered over 2 hours on Day -6 pre-HSCT. VP-16 60 mg/kg IV x 1 dose to be administered over 4 hours on Day -4.
  Radiation - administered at a rate of < 20 cGy/min in one of the following doses; 120 cGy/fraction are administered at no less than 4-hour intervals three times/day or 2 times/day for a total of 10 doses (1200 cGy) over 4 days (Day -8, -7, -6 and -5), or doses of 150 cGy/fraction twice daily for a total of 8 doses (1200 cGy) over 4 days (Day -8, -7, -6 and -5). VP-16 60 mg/kg IV x 1 dose to be administered over 4 hours on Day -4 pre-HSCT.
  Cyclophosphamide 100 mg/kg IV x 1 dose to be administered over 2 hours on Day -2 pre-HSCT. G-CSF 5 mcg/kg SQ or IV to start on Day +5 post-HSCT and continue until ANC > 500/mm3 x 3 days.
  Other Names: Etoposide and Carmustine; BCNU and VP-16
  Arms: Autologous Transplant
Drug: Non-myeloablative Conditioning regimen — Fludarabine 30 mg/m2 IV x 3 doses total to be administered daily over 30 minutes on Days -6, -5 and -4 pre-HSCT. Cyclophosphamide 750 mg/m IV x 3 doses total to be administered daily over 1 hour on Days -6, -5 and -4 pre-HSCT. Administer cyclophosphamide approximately 4 hours after start of fludarabine infusion. Rituximab 375 mg/m2 IV x 4 doses total to be administered on Days -13 and -6 pre HSCT and Days +1 and +8 post HSCT.
  Other Names: Fludarabine, Cyclophosphamide, and Rituximab; Fludara, Cytoxan®, and Rituxan
  Arms: Allogeneic Transplant
Procedure: Allogeneic transplant — Infusion of G-CSF mobilized allogeneic hematopoietic stem cells
  Other Names: HSCT
  Arms: Allogeneic Transplant
Procedure: Autologous transplant — Infusion of G-CSF mobilized autologous hematopoietic stem cells
  Other Names: HSCT
  Arms: Autologous Transplant
Drug: Rituximab maintenance therapy — Patients must have sufficiently recovered from autologous HSCT in order to receive rituximab maintenance therapy as specified below:
  Dose #1: Day +42 post-autologous HSCT Dose #2: Day +49 post-autologous HSCT Dose #3: Day +56 post-autologous HSCT Dose #4: Day +63 post-autologous HSCT
  Other Names: Rituxan
  Arms: Autologous Transplant
Drug: GVHD Prophylaxis — Tacrolimus 0.09 mg/kg/day PO, based on body weight formulas will start on Day -2 and continue until Day +90 post-HSCT. Tacrolimus (or cyclosporine, if applicable) will be given orally in a twice-daily divided dose. Methotrexate 5 mg/m2 Intravenous Pyelogram (IVP) will be administered on Days +1, +3 and +6 post-HSCT.
  Other Names: Tacrolimus and Methotrexate; Prograf® and MTX
  Arms: Allogeneic Transplant

SUMMARY:
This study is designed as a Phase II/III, multi-center trial, comparing two transplant strategies to determine whether non-myeloablative allogeneic Hematopoietic Stem Cell Transplantation (HSCT) will improve long-term progression-free survival compared to autologous HSCT. Recipients will be biologically assigned to the appropriate treatment arm depending on the availability of a Human Leukocyte Antigen (HLA) matched sibling.

DETAILED DESCRIPTION:
BACKGROUND:

Although patients with follicular non-Hodgkin's lymphoma (NHL) typically experience a relatively indolent course, the disease is rarely curable with conventional chemotherapy. Patients with follicular NHL are usually treated only when symptoms require palliation or if bulky disease exists since no survival advantage has been shown as compared to administering conventional treatment at initial diagnosis. While most patients achieve a remission with initial chemotherapy, a continuous pattern of relapse occurs, resulting in progressively shorter remission durations. Additionally, the increased response rates conferred by anthracycline-containing regimens have not translated into improved survival and thus the median survival time of 6 to 10 years has not been significantly impacted over the last decade.

DESIGN NARRATIVE:

The overall study design is a comparison of two treatment arms determined by biologic assignment, based on the availability of an HLA-matched sibling, in patients diagnosed with relapsed follicular non-Hodgkin's lymphoma. Patients without an HLA-matched sibling will receive an autologous HSCT. Patients with an HLA-matched sibling will receive a non-myeloablative allogeneic HSCT.

The overall study design is that of biologic assignment, based on the availability of an HLA-matched sibling, to one of two strategies to improve the outcome for follicular lymphoma patients with chemosensitive disease. All patients will undergo cytoreduction with cyclophosphamide 4 gm/m^2 and rituximab 375 mg/m^2 x 2 doses. Rituximab will be given in two doses, approximately 1 week apart, with the cyclophosphamide administered the day after the first dose of rituximab. Patients assigned to the autologous arm will have their hematopoietic stem cells mobilized from this cytoreductive regimen. Patients with an HLA-matched sibling will undergo a non-myeloablative allogeneic HSCT. Pre-transplant conditioning will consist of fludarabine 30 mg/m^2/day and cyclophosphamide 750 mg/m^2/day x 3 days with rituximab 375 mg/m^2/day on Days -13 and -6 pre-HSCT and on Days +1 and +8 post-HSCT. The immunosuppressive regimen will consist of tacrolimus and methotrexate (MTX) to control graft-versus-host and host-versus-graft reactions. Patients without an HLA-matched sibling who have collected an adequate autologous hematopoietic cell graft, defined as at least 2.0 * 10^6 CD34+ cells/kg, will receive a preparative regimen of total body irradiation (TBI) 1200 cGy or Carmustine (BCNU) 15 mg/kg. In addition, VP-16 60 mg/kg and cyclophosphamide 100 mg/kg will be given for both autologous preparative regimens. Post-autologous HSCT therapy with rituximab 375 mg/m^2 weekly x 4 doses will commence between Days 42-75 post-HSCT.

ELIGIBILITY:
Initial Patient Inclusion Criteria:

* Histologically confirmed recurrent Revised European American Lymphoma (REAL) classification follicle center lymphoma, follicular grades I and II, OR histologically confirmed World Health Organization (WHO) classification follicular lymphoma grades 1, 2, 3a or 3b; for either classification, the diffuse component or presence of large cleaved cells (if present) cannot be more than 50% of high power field; patients do not have to express t(14;18) to be eligible
* Received three or fewer prior regimens of chemotherapy; monoclonal antibody therapy and involved field radiation therapy will not be counted as a prior therapy
* Beyond first Complete Remission (CR) or first Partial Remission (PR) AND demonstrate chemosensitive disease; chemosensitive disease will be defined as less than 20% bone marrow involvement in the aspirate or core biopsy with follicular lymphoma AND lymph node size in axial diameter of less than 3 cm or a greater than 50% reduction in estimated lymph node volume to be measured as product of bi-dimensional measurements; Positron Emission Tomography (PET) scanning will not be used for staging or response purposes

  * Patients with adequate organ function as measured by:

    1. Cardiac: left ventricular ejection fraction at rest at least 45%
    2. Hepatic: bilirubin less than 2 times the upper limit of normal and alanine transaminase (ALT) and aspartate aminotransferase (AST) less than 3 times the upper limit of normal
    3. Renal: creatinine clearance greater than 40 mL/min
    4. Pulmonary: Diffusing capacity of the lung for carbon monoxide (DLCO), Forced expiratory volume in one second (FEV1), and Forced vital capacity (FVC) greater than 50% of predicted (corrected for hemoglobin)
  * If the patient is younger than 18 years of age and they have reached the age of assent, then they must have completed the local Institutional Review Board (IRB) assent process.
  * Able to receive cyclophosphamide and rituximab mobilization chemotherapy no earlier than 3 weeks from the beginning of the most recent cycle of salvage chemotherapy and no later than 6 weeks from enrollment

Patient Inclusion Criteria for Proceeding to Hematopoietic Stem Cell Transplant (HSCT):

* Collection of an autologous or allogeneic graft of at least 2.0 * 10^6 CD34+ cells/kg
* Blood count recovery defined as Absolute Neutrophil Count (ANC) greater than 1000/mm3 and platelets greater than 100 * 10^9/L

Patient Inclusion Criteria for Maintenance Therapy:

* Liver and renal function tests within the inclusion criteria for initial autograft
* Off intravenous antibiotics and off amphotericin B formulations for proven, probable or possible fungal infections
* No active Cytomegalovirus (CMV) infections or for patients with CMV infection post-autograft, treated with ganciclovir, valganciclovir, or foscarnet per institutional guidelines and CMV antigenemia negative
* Mucositis resolved and off hyperalimentation

Exclusion Criteria:

* Karnofsky performance score less than 70%
* Follicular lymphoma that show histologic evidence of transformation
* Uncontrolled hypertension
* Patients with uncontrolled bacterial, viral or fungal infection (currently taking medication and progression without clinical improvement).
* Prior malignancies except resected basal cell carcinoma or treated cervical carcinoma in situ; cancer treated with curative intent more than 5 years previously will be reviewed on a case-by-case basis by a Protocol Chair or Medical Monitor.
* Pregnant (positive Beta Human chorionic gonadotropin (β-HCG)) or breastfeeding
* Seropositive for Human immunodeficiency virus (HIV)
* Unwilling to use contraceptive techniques during treatment
* Prior autologous or allogeneic HSCT
* Known anaphylactic reaction to rituximab

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-08; Primary Completion 2006-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Horowitz, MD, Study Director — Center for International Blood and Marrow Transplant Research
Locations (30):
- United States (30):
  - City of Hope National Medical Center, Duarte, California
  - Scripps Clinic, La Jolla, California
  - UCSD Medical Center, La Jolla, California
  - Stanford Hospital and Clinics, Stanford, California
  - University of Florida College of Medicine (Shands), Gainesville, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - BMT Group of Georgia, Atlanta, Georgia
  - Loyola University, Atlanta, Georgia
  - Indiana BMT at Beech Grove, Beech Grove, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Karmanos Cancer Institute/BMT, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Kansas City Cancer Centers, Kansas City, Missouri
  - Washington University/Barnes Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals of Cleveland/Case Western, Cleveland, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Oregon Health Sciences University, Portland, Oregon
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas/MD Anderson CRC, Houston, Texas
  - Virginia Commonwealth University MCV Hospitals, Richmond, Virginia
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Tomblyn MR, Ewell M, Bredeson C, Kahl BS, Goodman SA, Horowitz MM, Vose JM, Negrin RS, Laport GG. Autologous versus reduced-intensity allogeneic hematopoietic cell transplantation for patients with chemosensitive follicular non-Hodgkin lymphoma beyond first complete response or first partial response. Biol Blood Marrow Transplant. 2011 Jul;17(7):1051-7. doi: 10.1016/j.bbmt.2010.11.004. Epub 2010 Nov 10. PMID 21073974

RESULTS

PARTICIPANT FLOW:
Groups:
- Autologous Hematopoietic Stem Cell Transplant (HSCT): Autologous HSCT preceded by bone marrow ablation including cyclophosphamide 100mg/kg, etoposide 60mg/kg and either radiation therapy at 1200cGy or carmustine at 15mg/kg
- Allogeneic Hematopoietic Stem Cell Transplant (HSCT): Human Leukocyte Antigen (HLA) matched sibling donor HSCT preceded by bone marrow ablation consisting of cyclophosphamide (750mg/m^2/day from day -6 to -4) fludarabine (30mg/m^2/day from day -6 to -4)
Period: Overall Study
Arm/Group | Autologous Hematopoietic Stem Cell Transplant (HSCT) | Allogeneic Hematopoietic Stem Cell Transplant (HSCT)
Started | 22 | 8
Completed | 15 | 7
Not Completed | 7 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Autologous Hematopoietic Stem Cell Transplant (HSCT) | Allogeneic Hematopoietic Stem Cell Transplant (HSCT) | Total
Number analyzed (Participants) | 22 | 8 | 30
Age, Continuous [Median (Full Range); unit: years] | 50 [36 to 66] | 48 [40 to 64] | 49 [36 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 3 | 15
  Male | 10 | 5 | 15
Region of Enrollment [Number; unit: participants]
  United States | 22 | 8 | 30
Disease Status at Enrollment [Number; unit: Participants]
  First Relapse | 2 | 0 | 2
  Second Relapse | 1 | 0 | 1
  Third Relapse | 1 | 0 | 1
  Second Partial Remission | 8 | 3 | 11
  Third Partial Remission | 3 | 1 | 4
  Second Complete Remission | 6 | 3 | 9
  Third Complete Remission | 1 | 1 | 2
Number of Prior Therapies [Median (Full Range); unit: Number of therapies] | 2 [1 to 3] | 2 [1 to 3] | 2 [1 to 3]
Months from diagnosis to transplant [Median (Full Range); unit: months] | 39.8 [9.8 to 110.5] | 28.9 [16.2 to 64.7] | 33.6 [9.8 to 110.5]

OUTCOME MEASURES:

1. Primary Outcome: Lymphoma Progression-free Survival
Time Frame: Three years post-Hematopoietic Stem Cell Transplant (HSCT)
Measure: Number; unit: participants
Arm/Group | Autologous Hematopoietic Stem Cell Transplant (HSCT) | Allogeneic Hematopoietic Stem Cell Transplant (HSCT)
Number analyzed (Participants) | 20 | 7
participants | 13 [43.8 to 89.6] | 6 [63.3 to 100]
Statistical Analysis 1: Comparison: Autologous Hematopoietic Stem Cell Transplant (HSCT); Test type: Superiority or Other; Kaplan-Meier Survival Probability = 62.7, 95% CI 2-sided [43.8 to 89.6]
Statistical Analysis 2: Comparison: Allogeneic Hematopoietic Stem Cell Transplant (HSCT); Test type: Superiority or Other; Kaplan-Meier Survival Probability = 85.7, 95% CI [63.3 to 100]

ADVERSE EVENTS:
Time Frame: 3-years post-transplant
Description: Serious adverse events are defined as events associated with death, life-threatening event, disability, congenital anomaly, required intervention to prevent permanent impairment or damage, hospitalization or other serious adverse event.
Arm/Group | Autologous Hematopoietic Stem Cell Transplant (HSCT) | Allogeneic Hematopoietic Stem Cell Transplant (HSCT)
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/7
Other Adverse Events (participants affected / at risk) | 0/20 | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autologous Hematopoietic Stem Cell Transplant (HSCT) (N=20) | Allogeneic Hematopoietic Stem Cell Transplant (HSCT) (N=7)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2006-01-17): https://cdn.clinicaltrials.gov/large-docs/60/NCT00096460/Prot_SAP_ICF_000.pdf